CLINICAL TRIAL: NCT04386317
Title: The Effect of A1- Adrenergic Receptor Antagonist Therapy on Cardiac and Striatal Transporter Uptake in Pre-Motor and Symptomatic Parkinson's Disease
Brief Title: Terazosin Effect on Cardiac Changes in Early Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michele Tagliati, MD, Professor and Vice Chairman, Director of Movement Disorders, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study#000540
Record Dates: First submitted 2020-04-24; First posted 2020-05-13 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: REM Sleep Behavior Disorder; Pre-motor Parkinson's Disease; Symptomatic Parkinson Disease
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease, Secondary | interventions — Terazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- terazosin therapy (Experimental): Daily oral doses of adrenergic blocker 5 mg or 10 mg. The dosage will be gradually increased from the initial recommended starting dose of 1 mg daily at bedtime and titrated stepwise to 2mg, 5mg or 10 mg weekly, according to patient tolerability, as measured by subjective complaints, arterial blood pressure and heart rate. The target dose will be 5 mg or 10 mg daily based on subject's tolerability.
  Interventions: Drug: Terazosin

INTERVENTIONS:
Drug: Terazosin — Fifteen patients with defined pre-motor PD risk and abnormal baseline 123I-MIBG uptake, with or without 123I-Ioflupane uptake abnormality or PD motor symptoms, will be recruited to receive daily oral doses of terazosin 5 mg or 10 mg. The dosage of terazosin will be gradually increased from the initial recommended starting dose of 1 mg daily at bedtime and titrated stepwise to 2mg, 5mg or 10 mg weekly, according to patient tolerability, as measured by subjective complaints, arterial blood pressure and heart rate. The target dose will be 5 mg or 10 mg daily based on subject's tolerability. Development of incompatibility will be addressed by individually adjusting the dose of terazosin.

SUMMARY:
Parkinson's disease (PD) is characterized by many non-motor symptoms that occur several years before the diagnosis, in particular idiopathic REM behavior disorder (iRBD), which is associated with autonomic impairment. The purpose of this study is to investigate the effect of treatment with the selective post-synaptic a1-adrenergic blocker terazosin on 123I-MIBG myocardial uptake in a population of subjects with defined pre-motor PD risks (i.e. hyposmia and RBD) and abnormal baseline 123I-MIBG uptake, with or without 123I-Ioflupane uptake abnormality or PD motor symptoms. Scintigraphic changes will be correlated to motor and non-motor severity of PD, measured by validated clinical scales and cardiac autonomic function tests.

DETAILED DESCRIPTION:
Based on the increased risk to develop PD, individuals with iRBD are currently considered ideal candidates for therapies that can possibly protects brain cells, due to the critical window of opportunity to intervene early before brain cell loss progresses significantly.

Early changes of PD are associated with a number of symptoms including loss of smell, constipation, anxiety and depression. In addition, early heart and brain abnormalities can be visualized using specialized imaging techniques called 123I-MIBG myocardial scintigraphy (MIBG) and dopamine transporter (DAT) single photon emission computerized tomography (SPECT) respectively. The combined presence of certain symptoms and the use of these imaging techniques are considered early markers of PD in individuals with iRBD.

In this study the investigators want to learn about the effect of treatment with the adrenergic blocker terazosin on MIBG abnormalities in iRBD patients at risk to develop PD. The investigators believe that reversing the MIBG abnormality might prelude to a slowing of the neurodegenerative process. This drug is approved by the U.S. Food and Drug Administration (FDA) for Benign Prostatic Hyperplasia (BPH) and Hypertension. However, terazosin is not approved by the FDA in patients with iRBD at risk for PD. The available doses for this drug oral formulations are 1mg, 2 mg, 5mg and 10 mg.

Changes visualized with the MIBG imaging technique will be correlated to the presence and severity of neurological (i.e. tremors, stiffness, slow movements, walking difficulties) and other symptoms associated with PD (i.e. abnormal smell, constipation, depression, color vision abnormalities), as measured by specific clinical scales and exams.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age between 50 and 85 years at time of enrollment.
* Diagnosis of idiopathic REM sleep behavior disorder (iRBD), established either as 'definite RBD' according to the criteria proposed by the International Classification of Sleep Disorders (ICSD)-2 [AASM, 2005] or 'probable RBD' following a score of 6 or higher in the RBD questionnaire (RBDSQ) [Nomura et al, 2011], with a score of at least 1 in subitems 6.1 to 6.4 of question 6 [Halsband et al, 2018].
* At least one of the following:

  1. Diagnosis of hyposmia, established as a University of Pennsylvania Smell Identification Test (UPSIT) score < 20th percentile for the individual's age group and sex.
  2. Functional constipation assessed by a scores > 4 on a questionnaire based on modified ROME IV diagnostic criteria.
  3. Color vision abnormality, as assessed using HRR Pseudoisochromatic Plates, in the absence of congenital dyschromatopsia
  4. Symptoms of depression, as assessed by a Beck Depression Inventory (BDI) fast screen score >3 or concurrent use of antidepressant medications.
* Abnormal 123I-MIBG myocardial scintigraphy, as defined by a Late H/M ratio < 2.2 and/or a WR >20%, with normal cardiac ejection fraction (LVEF >55%).
* Capacity to give informed consent

Exclusion Criteria:

* Secondary Parkinsonism, including tardive
* Concurrent dementia defined by a score lower than 22 on the MOCA
* Concurrent severe depression defined by a BDI fast screen score greater than 13
* Comorbidites related to SNS hyperactivity

  * Heart failure (LVEF< 45%)
  * Recent myocardial revascularization (< 12 weeks)
  * Hypertension (SBP >150 mmHg or DBP> 100mmHg)
  * Chronic Atrial fibrillation
  * Concurrent use of Alpha- adrenergic antagonist
  * Diabetes mellitus
  * COPD
  * Untreated Severe Sleep Apnea; Apnea-Hypopnea Index (AHI) > 30/h.
* Contraindication to the use of Terazosin

  * Recent myocardial infarction (< 48 h)
  * Ongoing angina pectoris
  * Cardiogenic shock or prolonged
  * Breast feeding
  * Current use of Phosphodiesterase type 5 inhibitors: sildenafil (Viagra TM), tadalafil (Cialis TM), or vardenafil (Levitra TM)
  * History of Priapism
  * Neurogenic orthostatic hypotensiondefiened as symptomatic decrease in BP> 20 mmHg systolic or > 10mmHg diastolic and HR increase < 20bpm on supine to sitting or standing
  * Blood pressure less than 110 mmHG systolic at screening or baseline visit
  * Use of investigational drugs whitin 30 days before screening
  * For female participant, Pregnacy, or plans for child-bearing during study period
* Allergy/hypersenstivity to iodine or study medication

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Differences in 123I-MIBG reuptake, as measured by early and late Heart to mediastinum (H/M) ratio, and Washout Ration (WR), at 26 weeks of treatment with the adrenergic blocker terazosin | At baseline and at 26 weeks after medication titration
  1) Differences in 123I-MIBG reuptake, as measured by early and late H/M ratio, and WR, at 26 weeks of treatment with the adrenergic blocker Terazosin.

SECONDARY OUTCOMES:
Incidence of adverse events | At baseline and at 26 weeks after medication titration
  Safety will be monitored collecting the type and frequency of adverse events, including clinical symptoms
Heart Rate variability changes from baseline at 26 weeks after study medication titration | At baseline and at 26 weeks after medication titration
  Beat-to-beat intervals will be registered to assess sympatho-vagal balance.
Incidence of abnormal vital signs | At baseline and at 26 weeks after medication titration
  Changes in vital signs (Blood pressure and Heart rate)

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Tagliati, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Michele L Lima Gregorio, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No